CLINICAL TRIAL: NCT06808412
Title: A Study on the Efficacy and Safety of Sintilimab Combined with Bevacizumab in Perioperative Neoadjuvant Chemotherapy for Locally Advanced Low Rectal Cancer
Brief Title: To Explore the Efficacy of Sintilimab Combined with Bevacizumab in Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: xiaohua li (Other)
Responsible Party: Sponsor-Investigator, xiaohua li, Associate Chief Physician, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20242241-C-1
Record Dates: First submitted 2025-01-20; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Rcctal Cancer
MeSH Terms: interventions — Bevacizumab; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with rectal cancer receiving sintilimab combined with bevacizumab and XELOX as a neoadjuvan (Experimental)
  Interventions: Drug: sintilimab combined with bevacizumab and XELOX

INTERVENTIONS:
Drug: sintilimab combined with bevacizumab and XELOX — Patients with locally advanced low rectal cancer receiving sintilimab combined with bevacizumab and XELOX as a neoadjuvant regimen during the perioperative period.

SUMMARY:
This is a prospective, exploratory clinical study. The primary endpoint of the study is to assess the pathological complete response (pCR) rate of tumors after neoadjuvant chemotherapy for rectal cancer using sintilimab combined with bevacizumab. The aim is to evaluate the efficacy and safety of sintilimab in combination with bevacizumab in the perioperative neoadjuvant chemotherapy for rectal cancer. The study includes two cohorts: Cohort A involves a retrospective collection of rectal cancer patients who previously received the XELOX regimen in the perioperative setting. Cohort B includes rectal cancer patients undergoing perioperative treatment with sintilimab and bevacizumab combined with XELOX as a neoadjuvant regimen.

Each of the trial group and historical control group requires 59 cases. The administration method for the trial group (Cohort B) is as follows:

Sintilimab: 200 mg, intravenous, Day 1, every 3 weeks. Bevacizumab: 7.5 mg/kg, intravenous, Day 1, every 3 weeks. Chemotherapy regimen: XELOX regimen.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A:

Rectal cancer patients who have previously received perioperative XELOX regimen treatment.

* Cohort B:

  1.Signed written informed consent prior to any trial-related procedures;

  2.Non-bedridden cases, regardless of gender, aged 18-75 years;

  3.Pathologically confirmed rectal adenocarcinoma, excluding anal squamous cell carcinoma;

  4.No prior antitumor treatment for rectal cancer. For those with Lynch syndrome, no antitumor treatment has been administered for the colorectal cancer related to this diagnosis;

  5.Based on high-resolution MRI, classified as T1-3bN1-2 or T3aN0 or T3bN0; no involvement of the levator ani muscle; negative mesorectal fascia (MRF) status; negative extramural vascular invasion (EMVI); no cancerous nodules;

  6.ECOG performance status of 0-1;

  7.Expected survival time > 3 months;

  8.Adequate organ function, with subjects meeting the following laboratory criteria:
  1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L without using granulocyte colony-stimulating factor in the past 14 days.
  2. Platelet count ≥ 100 x 10^9/L without transfusion in the past 14 days.
  3. Hemoglobin > 9 g/dL without transfusion or use of erythropoietin in the past 14 days;
  4. Total bilirubin ≤ 1.5 × upper limit of normal (ULN); if total bilirubin > 1.5 × ULN but direct bilirubin ≤ ULN, enrollment is also allowed;
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (patients with liver metastases are allowed if ALT or AST ≤ 5 × ULN);
  6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance (calculated by the Cockcroft-Gault formula) ≥ 60 ml/min;
  7. Good coagulation function, defined as an international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN;
  8. Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within normal range. If baseline TSH is outside the normal range, subjects can still be enrolled if total T3 (or FT3) and FT4 are within normal range;
  9. Normal levels of cardiac enzyme profile (subjects may still be enrolled if the investigator judges the laboratory abnormality to be of no clinical significance); (optional)

     9.For female subjects of childbearing potential, a urine or serum pregnancy test must be performed within 3 days prior to the first dose of the investigational drug (Day 1 of Cycle 1) with a negative result. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Non-childbearing potential females are defined as those who have been postmenopausal for at least one year, or have undergone surgical sterilization or hysterectomy;

     10.If there is a risk of conception, all subjects (regardless of gender) must use contraception with a failure rate of less than 1% throughout the treatment period and until 120 days after the last dose of the investigational drug (or 180 days after the last dose of chemotherapy).

     Exclusion Criteria:

     - 1. Diagnosed with malignant diseases other than rectal cancer within 5 years prior to the first administration (excluding cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or completely excised in situ carcinoma); 2.Currently participating in an interventional clinical study treatment, or received other investigational drugs or used investigational devices within 4 weeks prior to the first administration; 3.Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs, or drugs targeting another stimulus or co-inhibitory T cell receptors (including but not limited to CTLA-4, OX-40, CD137, etc.); 4.Received traditional Chinese medicine or immunomodulatory drugs with anti-tumor indications (including thymosin, interferon, interleukin, except for local use to control pleural effusion) within 2 weeks prior to the first administration.

     5.Experienced active autoimmune diseases requiring systemic treatment (e.g., use of disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years prior to the first administration. Alternative therapies (e.g., thyroid hormone, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatment;

     6.Receiving systemic glucocorticoid treatment within 7 days prior to the first administration of the study (excluding nasal, inhaled, or other forms of local glucocorticoids) or any other form of immunosuppressive therapy;

     Note: Physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are allowed;

     7.Presence of clinically uncontrollable abdominal effusion (patients who do not require drainage of effusion or who have not shown significant increase in effusion after stopping drainage for 3 days may be included);

     8.Known history of allogeneic organ transplantation (except for corneal transplantation) or allogeneic hematopoietic stem cell transplantation;

     9.Known allergy to the study drugs sintilimab, bevacizumab, or any active ingredients or excipients related to these investigational drugs;

     10.Presence of multiple factors affecting oral medication (e.g., inability to swallow, post-gastrointestinal resection, chronic diarrhea, and bowel obstruction);

     11.Not fully recovered from any toxicity and/or complications arising from any intervention prior to the start of treatment (i.e., ≤ grade 1 or return to baseline, excluding fatigue or hair loss);

     12.Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV 1/2 antibodies);

     13.Untreated active hepatitis B (defined as HBsAg positive with HBV-DNA copies exceeding the upper limit of normal for the testing laboratory at the study site);

     Note: Hepatitis B subjects meeting the following criteria may also be included:

     HBV viral load <1000 copies/ml (200 IU/ml) prior to the first administration; subjects should receive anti-HBV treatment throughout the study drug treatment period to prevent viral reactivation.

     Subjects with anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-) do not need to receive prophylactic anti-HBV treatment but require close monitoring for viral reactivation.

     14.Active HCV infection subjects (HCV antibody positive and HCV-RNA level above the lower limit of detection); 15.Received live vaccine within 30 days prior to the first administration (Cycle 1, Day 1); Note: Inactivated virus vaccine for seasonal influenza is allowed within 30 days prior to the first administration; however, intranasal live attenuated influenza vaccine is not permitted.

     16.Pregnant or breastfeeding women; 17.Presence of any severe or uncontrolled systemic diseases, such as:

  <!-- -->

  1. Significant abnormalities in rhythm, conduction, or morphology on resting ECG that are severe and symptomatic, such as complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmia, or atrial fibrillation;
  2. Unstable angina, congestive heart failure, chronic heart failure classified as NYHA class ≥ 2;
  3. History of any arterial thrombosis, embolism, or ischemia within 6 months prior to enrollment, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack;
  4. Poorly controlled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
  5. History of non-infectious pneumonia requiring glucocorticoid treatment within 1 year prior to the first administration, or current clinically active interstitial lung disease;
  6. Active pulmonary tuberculosis;
  7. Presence of active or uncontrolled infections requiring systemic treatment; Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
  8. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  9. Poorly controlled diabetes (fasting blood glucose (FBG) > 10 mmol/L); Urinalysis indicating urine protein ≥ ++, confirmed by 24-hour urine protein quantification > 1.0 g;
  10. Presence of mental disorders and inability to cooperate with treatment;
  11. Any history or evidence of disease that may interfere with study results, hinder subject participation throughout the study, abnormal treatment or laboratory test values, or other conditions deemed unsuitable for enrollment by the investigator due to potential risks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
assess the pathological complete response (pCR) rate of tumors after neoadjuvant chemotherapy for rectal cancer using sintilimab combined with bevacizumab | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cremolini C, Antoniotti C, Rossini D, Lonardi S, Loupakis F, Pietrantonio F, Bordonaro R, Latiano TP, Tamburini E, Santini D, Passardi A, Marmorino F, Grande R, Aprile G, Zaniboni A, Murgioni S, Granetto C, Buonadonna A, Moretto R, Corallo S, Cordio S, Antonuzzo L, Tomasello G, Masi G, Ronzoni M, Di Donato S, Carlomagno C, Clavarezza M, Ritorto G, Mambrini A, Roselli M, Cupini S, Mammoliti S, Fenocchio E, Corgna E, Zagonel V, Fontanini G, Ugolini C, Boni L, Falcone A; GONO Foundation Investigators. Upfront FOLFOXIRI plus bevacizumab and reintroduction after progression versus mFOLFOX6 plus bevacizumab followed by FOLFIRI plus bevacizumab in the treatment of patients with metastatic colorectal cancer (TRIBE2): a multicentre, open-label, phase 3, randomised, controlled trial. Lancet Oncol. 2020 Apr;21(4):497-507. doi: 10.1016/S1470-2045(19)30862-9. Epub 2020 Mar 9. PMID 32164906
- [Background] Gruenberger T, Bridgewater J, Chau I, Garcia Alfonso P, Rivoire M, Mudan S, Lasserre S, Hermann F, Waterkamp D, Adam R. Bevacizumab plus mFOLFOX-6 or FOLFOXIRI in patients with initially unresectable liver metastases from colorectal cancer: the OLIVIA multinational randomised phase II trial. Ann Oncol. 2015 Apr;26(4):702-708. doi: 10.1093/annonc/mdu580. Epub 2014 Dec 23. PMID 25538173
- [Background] Giantonio BJ, Catalano PJ, Meropol NJ, O'Dwyer PJ, Mitchell EP, Alberts SR, Schwartz MA, Benson AB 3rd; Eastern Cooperative Oncology Group Study E3200. Bevacizumab in combination with oxaliplatin, fluorouracil, and leucovorin (FOLFOX4) for previously treated metastatic colorectal cancer: results from the Eastern Cooperative Oncology Group Study E3200. J Clin Oncol. 2007 Apr 20;25(12):1539-44. doi: 10.1200/JCO.2006.09.6305. PMID 17442997
- [Background] Van Cutsem E, Rivera F, Berry S, Kretzschmar A, Michael M, DiBartolomeo M, Mazier MA, Canon JL, Georgoulias V, Peeters M, Bridgewater J, Cunningham D; First BEAT investigators. Safety and efficacy of first-line bevacizumab with FOLFOX, XELOX, FOLFIRI and fluoropyrimidines in metastatic colorectal cancer: the BEAT study. Ann Oncol. 2009 Nov;20(11):1842-7. doi: 10.1093/annonc/mdp233. Epub 2009 Apr 30. PMID 19406901
- [Background] Kabbinavar FF, Hambleton J, Mass RD, Hurwitz HI, Bergsland E, Sarkar S. Combined analysis of efficacy: the addition of bevacizumab to fluorouracil/leucovorin improves survival for patients with metastatic colorectal cancer. J Clin Oncol. 2005 Jun 1;23(16):3706-12. doi: 10.1200/JCO.2005.00.232. Epub 2005 May 2. PMID 15867200
- [Background] Chen G, Jin Y, Guan WL, Zhang RX, Xiao WW, Cai PQ, Liu M, Lin JZ, Wang FL, Li C, Quan TT, Xi SY, Zhang HZ, Pan ZZ, Wang F, Xu RH. Neoadjuvant PD-1 blockade with sintilimab in mismatch-repair deficient, locally advanced rectal cancer: an open-label, single-centre phase 2 study. Lancet Gastroenterol Hepatol. 2023 May;8(5):422-431. doi: 10.1016/S2468-1253(22)00439-3. Epub 2023 Mar 1. PMID 36870360
- [Background] Wang F, Jin Y, Wang M, Luo HY, Fang WJ, Wang YN, Chen YX, Huang RJ, Guan WL, Li JB, Li YH, Wang FH, Hu XH, Zhang YQ, Qiu MZ, Liu LL, Wang ZX, Ren C, Wang DS, Zhang DS, Wang ZQ, Liao WT, Tian L, Zhao Q, Xu RH. Combined anti-PD-1, HDAC inhibitor and anti-VEGF for MSS/pMMR colorectal cancer: a randomized phase 2 trial. Nat Med. 2024 Apr;30(4):1035-1043. doi: 10.1038/s41591-024-02813-1. Epub 2024 Mar 4. PMID 38438735
- [Background] Xu J, Jiang H, Pan Y, Gu K, Cang S, Han L, Shu Y, Li J, Zhao J, Pan H, Luo S, Qin Y, Guo Q, Bai Y, Ling Y, Yang J, Yan Z, Yang L, Tang Y, He Y, Zhang L, Liang X, Niu Z, Zhang J, Mao Y, Guo Y, Peng B, Li Z, Liu Y, Wang Y, Zhou H; ORIENT-16 Investigators. Sintilimab Plus Chemotherapy for Unresectable Gastric or Gastroesophageal Junction Cancer: The ORIENT-16 Randomized Clinical Trial. JAMA. 2023 Dec 5;330(21):2064-2074. doi: 10.1001/jama.2023.19918. PMID 38051328
- [Background] Molinari C, Passardi A. Why is neoadjuvant chemoradiation therapy underused for locally advanced rectal cancer? Expert Rev Gastroenterol Hepatol. 2016 Dec;10(12):1317-1319. doi: 10.1080/17474124.2016.1246182. Epub 2016 Oct 19. No abstract available. PMID 27754713
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342